CLINICAL TRIAL: NCT06534775
Title: PABLOS 2.0 - Chronic Pain After Sternotomy, Prospective Non-interventional Study
Brief Title: PABLOS 2.0 - Chronic Pain After Sternotomy
Acronym: PABLOS2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC24_0179
Record Dates: First submitted 2024-07-24; First posted 2024-08-02 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnary — The patients were included in a previous study (PABLOS) - These patients received locoregional anesthesia (LRA) by deep parasternal intercostal block (Deep-PIP) or bilateral superficial parasternal intercostal block (Superficial-PIP), compared with standard management (general anesthesia without LRA) for chronic postoperative pain after cardiac surgery by sternotomy.
  In PABLOS 2.0 study, the evaluation focuses on the presence of chronic pain between 12 and 24 months postoperatively. There is no intervention in PABLOS 2.0 study but only a questionnary.

SUMMARY:
The PABLOS study (NCT05345639) recently realised at the University Hospital of Angers looked at the place of loco-regional anesthesia (LRA) in the optimization of analgesia and the early post-operative recovery of patients operated from cardiac surgery by sternotomy.

All randomized patients (n=253) were followed for 30 days as part of PABLOS monitoring with the aim of optimizing acute care.

However, sternotomy surgery causes chronic pain with neuropathic components. Indeed, numerous recent studies suggest that cardiac surgery by median sternotomy is associated with the development of chronic sternal pain with an incidence of 11% to 56% one year after surgery. Most patients with chronic post-sternotomies pain report mild pain (1 to 3 on the Numerical Scale), however, up to 18% report moderate to severe pain (4 to 10 on the EN).

It therefore seems important to the investigator to evaluate the prevalence of chronic post-sternotomies pain within our PABLOS cohort and to know whether performing a post-operative LRA limits their occurrence.

DETAILED DESCRIPTION:
PABLOS 2.0 is a non-interventional cohort study with prospective data collection by telephone questionnary, with three groups from a single-center superiority interventional study. Patients remained blinded for the duration of the study.

The patients in the cohort come from the precedent PABLOS study (NCT05345639). They receive oral and written information, and confirm orally their non-opposition to participating in the PABLOS 2.0 study.

The specific procedures of the PABLOS 2.0 study are the collection using a telephone questionnary of the score of the numerical scale (from 0 to 10) of pain at rest and with effort, of the DN4 (proportion of chronic pain with a neuropathic component), of the EQ-5D-5L scale (quality of life) and of consumption of painkillers.

ELIGIBILITY:
Inclusion Criteria:

* Patient who participated in the PABLOS study (See below);
* French-speaking patient, able to understand and answer a questionnary

Exclusion Criteria:

* Patient who has had an operation for cardiac or thoracic surgery, including a REDUX (surgical revision) of sternotomy since their inclusion in the PABLOS study;
* Patient opposing the research.

PABLOS criteria (NCT05345639) :

Pre-inclusion criteria

* Adult patient (≥18 years old);
* Patient having planned cardiac surgery with performance of a sternotomy at the Angers University Hospital;
* Patient having signed consent;
* French-speaking patient, able to understand and answer a questionnary;
* Patient affiliated to or beneficiary of a social security scheme;

Criteria for confirming inclusion

* Hemodynamic stability at the end of surgical intervention;
* Absence of bleeding justifying immediate surgical revision

Non-inclusion criteria

* Known hypersensitivity to local anesthetics with amide bonds;
* Operation for cardiac surgical revision, including REDUX (surgical revision) of sternotomy;
* Emergency surgery;
* Surgery in a septic context (Endocarditis, Intravascular device infection);
* Weight less than 30kg;
* Severe psychiatric or cognitive disorder hindering assessment by questionnary;
* Pregnant, breastfeeding or parturient woman;
* Person deprived of liberty by judicial or administrative decision;
* Person subject to psychiatric care under duress;
* Person subject to a legal protection measure;
* Inclusion in another interventional study modifying post-operative pain management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the PABLOS study, without non-inclusion criteria, are pre-selected to participate in the study. These are patients from the original PABLOS study who underwent thoracic surgery by sternotomy at the Angers University Hospital. The PABLOS inclusion period extended from August 1, 2022 to August 2, 2023.
  Patients receive an information letter at home, containing all the information relating to the PABLOS 2.0 study, a few weeks before receiving a telephone call, as well as a booklet containing the questionnary. From this stage, the patient has the possibility of contacting the team to express their opposition to participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 253 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-08-18 (Estimated); Study Completion 2025-08-18 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of LRA | 12 to 24 months
  The main objective is to compare the effectiveness of LRA (bilateral transverse thoracic block or bilateral parasternal block) compared to standard management (general anesthesia without LRA) on late postoperative recovery after surgery heart by sternotomy.
  The main endpoint is defined by the presence at the time of the call of pain that has been evolving for > 3 months with a numerical scale >0. Self-assessment by numerical scale varies from 0 to 10 :
  * 0 being no pain
  * from 1 to 3 : mild pain
  * from 4 to 6 : moderate pain
  * from 7 to 10 : severe pain

SECONDARY OUTCOMES:
LRA Impact on the intensity of exercise pain | 12 to 24 months
  Exercise-induced pain self-assessed using a numerical scale ranging : 0, no pain, to 10, the maximum pain imaginable.(12 to 24 months depending on the date the interview was carried out) Pain location is taken into account : main location of the pain in predefined areas (back, head, thorax, saphenous harvest scar, abdomen)
LRA Impact on the prevalence of neuropathic pain | 12 to 24 months
  Evaluate by the DN4 questionnary assessement. The patient must answer 10 questions divided into 4 items. If the patient's score is equal to or higher than 4/10, the test is positive.
LRA Impact on daily consumption of analgesics | 12 to 24 months
  Evaluate by measurement of daily consumption of painkillers
LRA Impact on quality of life | 12 to 24 months
  Quality of life measured using the EQ-5D-5L score.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression Each dimension have five response levels: no problems (score 1), slight problems, moderate problems, severe problems and extreme problems (score 5).
  Higher scores mean a worse outcome
  Responses are coded as single-digit numbers expressing the severity level selected in each dimension.
To describe all-cause mortality in cardiac surgery patients | 12 to 24 months
  Measurement of prevalence of deaths since the end of PABLOS follow-up
Infection of the puncture point(s) event in context of LRA in the long term. | 12 to 24 months
  During the telephone call, investigator will ask the patient if he/she has had an infection of the puncture site(s) after the initial PABLOS follow-up period (i.e. after 30 days post-operatively).
sternotomy scar revision in context of LRA in the long term. | 12 to 24 months
  During the telephone call, investigator will ask the patient if he/she has the need for sternotomy scar revision after the initial PABLOS follow-up period (i.e. after 30 days post-operatively).

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Achille DEMARQUETTE, Angers, Maine Et Loire, France